CLINICAL TRIAL: NCT05088096
Title: Translation, Cultural Adaptation and Psychometric Properties of Urdu Version of Upper Limb Functional Index Questionnaire in Patients With Upper Limb Musculoskeletal Disorders
Status: Completed | Type: Observational
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Other Study IDs: UOL 0676
Record Dates: First submitted 2021-10-09; First posted 2021-10-21 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Upper Limb Nerve Lesion; Reliability; Validity
Keywords: Translation; Musculoskeletal injury; Upper limb

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A reliability and validity study for the cross culturally adapted and translated version of Upper limb musculoskeletal index questionnaire into Urdu language. This can be used for the reporting of upper limb musculoskeletal disorders including hand, shoulder and arm pathologies, carpel tunnel syndrome, osteoarthritis etc.

DETAILED DESCRIPTION:
Upper limb functional disorders are quite common among Pakistani population due to high demands of work either manual or using technologies, so these disorders are also of great matter of interest. Therefore, for evaluations, diagnosis and for better treatment, a subjective questionnaire is required and hence, ULFI is a commonly used outcome measure for upper limb.

It has been previously translated into many languages i.e. in native languages of respective countries for better understanding.

Upper limb functional index (ULFI) is originally in English language and much of the Pakistani population is Urdu speaking. That is why it is required to translate the ULFI questionnaire in Urdu language.

Translation guidelines from Beaton and colleagues followed. The patients with upper limb musculoskeletal disorders will be recruited.

Data collection procedure started after the approval from institution review board committee with reference no. IRB-UOL-FAHS/882/2021. Data were collected from the patients after taking consent from them. Data collected on their first visit and second reading taken after 1 week, after that treatment will be given.

Data Analysis:

Reliability:

The ULFI-Urdu will be applied two times by a physiotherapist to determine test-retest reliability. On the first day of assessment the physiotherapist will collect demographic data and patients will answer ULFI-Urdu. For intra-rater reliability, ULFI-Urdu will be reapplied 48 hours later. Between two assessments, no treatment will be provided to minimize clinical differences. The first visit of the patient will be comprised of complete assessment along with the completion of outcome measures and upon his/her second visit the patient outcome measures will be completed before giving any treatment.

Validity:

Construct validity will be assessed by determining pearson correlation between ULFI-Urdu and DASH, ULFI-Ur and SF-12 Ur questionnaire.

Statistical Analysis:

The Kaiser-Meyer-Olkin measure of sampling adequacy will be used to assess for factor analysis and the Barlett test of sphericity, to ensure sampling adequacy. Reliability will be assessed with Cronbach alpha, split half test and test-retest method. Floor and ceiling effects will be determined by calculating the rate of participants that obtained the lowest (0) or highest (80) scores and will be considered present if more than 15 % of the participants achieved the highest or lowest score. Validity will be assessed by explanatory factorial analysis of the ULFI scores obtained at the first meeting. Principal components analysis will be performed with varimax rotation if it will be necessary. The number of potential factors will be suggested by scree plot, Eugen value cut-off >1.0, and 10 % variance. Convergent and divergent validity will be assessed with correlation between pain at rest, activity, DASH score, stiffness, physical function, total score and ULFI score.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients will be included.
* Sub-acute or chronic conditions of upper limb musculoskeletal disorders.
* Musculoskeletal disorders such as carpal tunnel syndrome (CTS), tendonitis or tenosynovitis, osteoarthritis, cramp of the hand or forearm from prolonged periods of repetitive movement, hand-arm vibration syndrome (HAVS).
* Patients with unilateral disorders will be included.

Exclusion Criteria:

* Presence of other significant rheumatic disease variants.
* Severe inflammatory arthritis as confirmed by physical examination.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects with upper limb musculoskeletal disorders will be enrolled in the study with age limits from 18-40 years. Data will be entered for the first and then after a duration of few days for reliability and validity of questionairre.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Cross cultural adaptation, translation, reliability and validity of Upper limb functional Index in patients with musculoskeletal disorders | 1 week
  Upper limb musculoskeletal disorder index will be translated into Urdu and will be cross culturally adapt throughout.
Cross cultural adaptation, translation, reliability and validity of Upper limb functional index (ULFI) | 1 week
  It will be assessed for reliability and validity.

CONTACTS AND LOCATIONS:
Overall Officials: Fareeha Amjad, Study Director — University of Lahore
Locations (1):
- Ayesha Arooj, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arooj A, Amjad F, Tanveer F, Arslan AU, Ahmad A, Gilani SA. Translation, cross-cultural adaptation and psychometric properties of Urdu version of upper limb functional index; a validity and reliability study. BMC Musculoskelet Disord. 2022 Jul 20;23(1):691. doi: 10.1186/s12891-022-05628-8. PMID 35858863